CLINICAL TRIAL: NCT07063524
Title: Principle Investigator
Brief Title: Transcutaneous Electrical Stimulation and Controlled Heat in People With and Without Diabetes
Acronym: TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Responsible Party: Principal Investigator, Massood Atashbar, PI, Western Michigan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201131
Record Dates: First submitted 2024-05-10; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diabetes; Heat; Perfusion; Complications
MeSH Terms: conditions — Diabetes Mellitus | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Pilot study of a single group of people with and without diabetes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Blood perfusion (Experimental): Blood flow at the foot with the application of heat and electrical stimulation
  Interventions: Device: Electrical stimulation

INTERVENTIONS:
Device: Electrical stimulation — Electrical stimulation with controlled heat during the intervention
  Other Names: controlled heat

SUMMARY:
The investigators would like to see if the combination of TENS and controlled heat in a boot increases blood flow to the foot more than baseline or heat alone in people with and without diabetes. This may help people with diabetes and a diabetic wound that will not heal.

DETAILED DESCRIPTION:
Procedure

1. Sit comfortably in a reclining chair for 5 minutes while temperature, SPO2, and heart rate are taken, and any further questions can be answered with a pulse oximeter and temperature

   a. The procedure for temperature, heart rate, and blood saturation rate will be taken using a Homedics Non-Contact Infrared Thermometer. The infrared beam will be pointed at the subject's forehead at approximately 1 foot away, and within 2 seconds, the temperature will be recorded and time-stamped.

   b. Procedure for the Pulse Oximeter- A SPO2 Pulse Oximeter will be placed on the subject's foot. The SPO2 sensors are embedded in the insole. The oxygen saturation level and pulse rate will be documented. The pulse oximeter will be cleaned with isopropyl alcohol before and after each use.
2. Temperature

   a. The procedure for taking Room temperature-Reading of the room temperature via the thermostat located in the lab.
3. Once the baseline temperature, SPO2, heart rate, and room temperature are documented, a PPG sensor will be located and embedded in the insole.

   a. Procedure for a PPG sensor- A PPG sensor is very similar to the pulse oximeter on the finger. The PPG also works on infrared light, similar to the pulse oximeter, and will data collection throughout the experiment.
4. 5-min of blood perfusion will be recorded at the dominant leg/foot.

   a. Procedure for recording blood perfusion- Once the subject's foot is on the insole, recordings of blood perfusion can be made from software. The PPG sensor will have a lead wire that connects to a USB port from the PPG to the computer for the data.
5. A boot will be placed on the patient's dominant leg with the subject still sitting; once comfortable with the boot, 5-more minutes of blood perfusion will be measured

   a. Procedure for putting on the boot- This boot is commercially available. The subject will put their foot into a padded insole, and straps will secure the foot and portion that goes up to the knee (picture below). The straps can be fastened to the subject comfort. It should not feel too tight or uncomfortable.
6. After 5 minutes of just the boot, the controlled heat in the boot will be turned on, and blood perfusion will be measured for 5 minutes. The heat will never be higher than 36-38 degrees C.

   a. Procedure for using controlled heat in the boot-With in the boot, five thermistors emit heat and are designed to increase heat. Once the heat is turned on, warmth will be felt at the subject foot and leg. The subjects and PI can see a digital readout of the heat on the computer screen. The temperature will not go higher than 38 deg C and be kept in the 36-38 deg C range. Past research has shown that this is a comfortable and safe approach.6-9 But the subjects are in full control of the heat, and the investigators can turn it down if it feels too warm.
7. After 5 minutes of heat, electrical stimulation will be added. It will be turned to an intensity that is comfortable to the subject but not high enough for a muscle contraction. The intensity will never be higher than 20 milliamps.

   a. Procedure for Electrical stimulation- An electrical stimulator with non-adhesive electrodes embedded in the insole will be used. 4-electrodes will be activated at the insole at the bottom of the foot. The electrodes are connected to an electrical stimulator. The intensity of the stimulus will never be high enough to cause a muscle contraction and be uncomfortable for the subject. The subject will be asked if they are comfortable and given the option to decrease or increase the stimulus (throughout the data collection). The intensity will never be over 20 mA.
8. This combination of electrical stimulation and heat will last 30 minutes while blood perfusion is measured.

   a. The procedure of controlled heat and electrical stimulation software will measure both the input of the heat and electrical stimulation, with the safety of the controlled heat, which will never go above 38 degrees C. The subject will always control the electrical stimulation and never experience any discomfort. The subject should not feel any muscle contraction or go over 20 milliamps with the intensity.
9. After 30 minutes, all elements will be turned off, and a final measurement will be made for 10-min.

   1. Recording blood perfusion with electrical stimulation and heat. The electrical stimulation and heat units will be turned off, but the PPG sensors located in the insole will collect blood perfusion readings while the subjects are sitting in a chair.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged between 45-75 years old
* Clinical diagnosis of Type I or Type II diabetes
* Controlled diabetes mellitus (HbA1c ≤ 7%)

Exclusion Criteria:

* Pregnancy
* Current smoker
* Diagnosed neuropathy
* Uncontrolled hypertension (HTN)
* Allergy to tape or electrodes
* Diagnosis of dementia
* History of knee joint replacement
* Significant joint pain (e.g., back, hip, or ankle) that may limit the ability to wear a boot for 60 minutes
* Contraindications to TENS, including:

  * Presence of pacemakers
  * Dermatological conditions
  * Abnormal sensation in the knees
* Severe medical or neurological conditions, including:

  * Chronic obstructive pulmonary disease
  * Cardiovascular disease
  * Arteriosclerosis obliterans
  * Cerebrovascular accident
  * Lumbar disc disorders (e.g., herniation)
  * Rheumatoid arthritis
* Fear of electrical stimulation

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood Perfusion | During 30 minutes of electrical stimulation and heat application.
  Peripheral Blood Perfusion and Oxygen Saturation (SpO₂) assessed using pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Massood Atashbar, PhD, Principal Investigator — Western Michigan University
Locations (1):
- Western Michigan University, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No